CLINICAL TRIAL: NCT00711048
Title: A Phase I, Two Centre, Double-blind, Randomized, Cross-over Study to Evaluate AZD1386 in Single Doses of 30 mg and 95 mg Compared to Placebo in a Multimodal Experimental Pain Model on Esophageal Sensitivity and Development of Sensitization in Healthy Male Volunteers
Brief Title: Esophageal Hypersensitivity Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Berner Hansen, MD, PhD, Acting Medical Science Director, Emerging Products CV/GI, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D9127C00001; 2008-000313-30
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Pain; Esophageal Sensitivity
Keywords: GERD; healthy volunteer; esophagus; pain
MeSH Terms: conditions — Pain; Gastroesophageal Reflux | interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 30 mg, oral, single dose
  Interventions: Drug: AZD1386
- 2 (Experimental): 95 mg, oral, single dose
  Interventions: Drug: AZD1386
- 3 (Placebo Comparator): Oral solution, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — oral, single dose
  Arms: 1; 2
Drug: Placebo — Oral solution, single dose
  Arms: 3

SUMMARY:
The purpose of the study is to compare sensitivity and sensitization of visceral pain in the esophagus using different pain stimuli

ELIGIBILITY:
Inclusion Criteria:

* Provision of written consent
* Clinically normal physical findings
* Sensitization potential

Exclusion Criteria:

* Clinically significant illness within 2 weeks prior to the first dose of investigational product
* History of clinically significant disease
* Use of prescribed medication during the 2 weeks before administration of the first dose of investigational product

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-06; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
VAS scale and clock | Several occasions during the study days

SECONDARY OUTCOMES:
VAS scale and pressure, VAS scale and current, VAS scale and acid volume | Several occasions during the study days
Pharmacokinetic variables | Several occasions during the study days
Safety variables (adverse events, blood pressure, safety lab, ECG and body temperature) | Several occasions during the study days

CONTACTS AND LOCATIONS:
Overall Officials: Marie Sundin, Study Director — AstraZeneca R&D, Mölndal, Sweden; Peter Funch-Jensen, MD, PhD, Principal Investigator — Aarhus University Hospital, Dept of Surgical Gastroenterology, Aarhus, Denmark
Locations (2):
- Research Site, Aarhus, Denmark
- Research Site, Gothenburg, Sweden

REFERENCES:
- [Derived] Krarup AL, Ny L, Astrand M, Bajor A, Hvid-Jensen F, Hansen MB, Simren M, Funch-Jensen P, Drewes AM. Randomised clinical trial: the efficacy of a transient receptor potential vanilloid 1 antagonist AZD1386 in human oesophageal pain. Aliment Pharmacol Ther. 2011 May;33(10):1113-22. doi: 10.1111/j.1365-2036.2011.04629.x. Epub 2011 Mar 16. PMID 21410733